CLINICAL TRIAL: NCT02437123
Title: The Cedar Project: Impact of mHealth for HIV Prevention Among Young Indigenous People Who Use Illicit Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H13-02718
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2016-07

CONDITIONS: Drug Addiction; HIV
Keywords: mHealth; Indigenous; HIV prevention; substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Cedar Project mHealth Intervention (Experimental): The Cedar Project mHealth intervention consists of a package of culturally-safe supports, including a mobile phone and long-distance cellular plan, weekly two-way text messaging, and support from community-based Cedar Advocates.
  Interventions: Behavioral: The Cedar Project mHealth intervention
- Comparison group (No Intervention): The comparison group will be sampled from The Cedar Project, an ongoing cohort study of young Indigenous people who use drugs under its existing informed consent with no change whatsoever to their participation in the overall study.

INTERVENTIONS:
Behavioral: The Cedar Project mHealth intervention
  Arms: The Cedar Project mHealth Intervention

SUMMARY:
This study will examine the effect of a culturally-safe two-way supportive text message intervention to reduce HIV vulnerability among young Indigenous people who use illicit drugs in a community-based setting.

The study is nested within The Cedar Project, an ongoing cohort study addressing HIV and Hepatitis C vulnerability among young Indigenous people who use drugs in Vancouver and Prince George, British Columbia, Canada. Indigenous collaborators and investigators, collectively known as the Cedar Project Partnership, govern the entire research process.

A stratified Zelen pre-randomized design will be used to identify a random selection of cohort members to be offered the Cedar Project mHealth intervention with consent. Participants in the intervention arm will receive a package of supports, including a mobile phone and long-distance plan, weekly two-way supportive text messaging via the WelTel platform, and support from Cedar Advocates. Those drawn from the cohort study population as the comparison group will continue on in the usual Cedar Project study under its existing informed consent with no change whatsoever to their participation in the overall study.

The main outcome is an HIV propensity score, assessed at six months and one year. Secondary outcomes include HIV risk, resilience, access to drug-related services, psychological distress, and connection to culture measured at six months and one year. Primary analysis is by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled in the Cedar Project
* completed main Cedar Project Baseline questionnaire and attended at least one follow-up visit since 2009
* had not tested positive for HIV
* joined study in Vancouver or Prince George
* alive at initiation of Cedar Project mHealth study

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
HIV propensity score | 0, 6 and 12 months
  Previous analyses of Cedar Project data have identified several factors as associated with HIV infection. These will be used to build a propensity score for HIV risk. Change in this score from baseline will be used to determine the impact of the intervention on HIV vulnerability over the prior six-month period.

SECONDARY OUTCOMES:
HIV risk | 0, 6 and 12 months
  Several self-reported binary measures will be used to determine the impact of the intervention on HIV risk in the prior six month period, including: recent injection drug use, high frequency drug use, needle sharing, and participation in sex work.
Resilience | 0, 6 and 12 months
  Resilience, or the ability to cope with stress in the face of adversity, will be characterized using the Connor-Davidson Resilience Scale (CD-RISC). The CD-RISC scale measures resilience via 25 items on a 5-point scale with scores ranging between 0-100, with higher scores indicating greater resilience.
Access to drug-related services | 0, 6 and 12 months
  Self-reported access to drug-related services, including opioid substitution therapy, needle exchange, safe injection facility, and drug treatment in the previous six month period will be ascertained from the main Cedar Project questionnaire. Proportions of participants reporting access to these services will be compared in the intervention and control groups. We will also determine if there are differences among treated and control groups in terms of proportion of people who tried to quit in the previous six-month period.
Connection to culture | 0, 6 and 12 months
  Connection to Indigenous culture has been hypothesized as a key protective factor for young Indigenous people who use drugs. It will be assessed using two dichotomous variables that measure cultural activity in the prior six-month period including: (1) Self-reported participation in traditional ceremonies (including: potlatch, feast, fast, burning ceremony, washing ceremony, naming ceremony, big/smoke house, rights of passage, smudge, dances, or any other traditional Indigenous ceremony); (2) frequently living by traditional culture (never/rarely vs. often/always). These variables were defined by Earl Henderson (Cree-Métis) and Violet Bozoki (Lheidli T'enneh Nation) who are Indigenous Elders, traditional knowledge keepers, and members of the Cedar Project Partnership.
Psychological distress | 0, 6 and 12 months
  The Symptom Checklist-90-R (SCL-90-R) is a 90-item self-reported symptom inventory that measures the severity of nine dimensions of psychological distress in the past three months scored on a five-point Likert scale (from not at all to extremely). Participants' SCL-90-R scores will be transformed into an average Global Severity Index ranging between 0-1.5, providing a single average measure that profiles overall degree of psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Health Evaluation and Outcome Sciences, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Jongbloed K, Friedman AJ, Pearce ME, Van Der Kop ML, Thomas V, Demerais L, Pooyak S, Schechter MT, Lester RT, Spittal PM; Cedar Project Partnership. The Cedar Project WelTel mHealth intervention for HIV prevention in young Indigenous people who use illicit drugs: study protocol for a randomized controlled trial. Trials. 2016 Mar 9;17(1):128. doi: 10.1186/s13063-016-1250-3. PMID 26957103